CLINICAL TRIAL: NCT03322085
Title: The Influence of Catheter Ablation for Atrial Fibrillation on Atrial Electrical Remodeling and the Relationship Between Electrical Remodeling and Structural Remodeling
Brief Title: The Influence of Catheter Ablation for Atrial Fibrillation on Atrial Electrical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Ruiqin xie, director of cardiology department, The Second Hospital of Hebei Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xierqdoctorER
Record Dates: First submitted 2017-09-28; First posted 2017-10-26 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; atrial electrical remodeling
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- paroxysmal AF with radiofrequency ablation (Experimental): radiofrequency catheter ablation therapy
  Interventions: Procedure: radiofrequency ablation or cryoballoon
- persistent AF with radiofrequency ablation group (Experimental): radiofrequency catheter ablation therapy
  Interventions: Procedure: radiofrequency ablation or cryoballoon
- paroxysmal AF with cryoballoon group (Experimental): cryoballoon ablation therapy
  Interventions: Procedure: radiofrequency ablation or cryoballoon

INTERVENTIONS:
Procedure: radiofrequency ablation or cryoballoon — Patients in radiofrequency ablation group receive circumferential pulmonary vein isolation,and no additional ablation is performed in the extrapulmonary sites unless the patient is diagnosed with atrial flutter before the operation. And Cryoablation is performed using a single cryoballoon. The diameter of the cryoballoon is determined as 28 mm or 23 mm according to pulmonary venography results.

SUMMARY:
This study explored the influence of radiofrequency catheter ablation and cryoballoon ablation on atrial electrical remodeling in patients with atrial fibrillation,the relationship between atrial electrical remodeling and structural remodeling,and which indicators are associated with atrial recurrence after catheter ablation.

DETAILED DESCRIPTION:
From September 2017 to September 2019, the investigators enroll consecutive patients with symptomatic atrial fibrillation (AF) who were scheduled for an initial catheter ablation, including paroxysmal and persistent AF.Patients are divided in to three group: paroxysmal AF in radiofrequency ablation group, persistent AF in radiofrequency ablation group, and paroxysmal AF in Cryoablation group.

1. Paroxysmal AF group: The p-wave duration, P wave dispersion and P wave amplitude are detected before and 24 hours after procedure.The atrial effective refractory period, refractory period dispersion, frequency adaptation and atrial conduction time were tested before and after procedure. Detect atrial electromechanical conduction time in the tissue doppler before and 1 week after procedure.
2. Persistent AF group: The p-wave duration, P wave dispersion and P wave amplitude are detected 24 hours after procedure.The atrial effective refractory period, refractory period dispersion, frequency adaptation and atrial conduction time were tested after procedure. Detect atrial electromechanical conduction time in the tissue doppler 1 week after procedure.
3. Method of detection of atrial electrical remodeling: 1). the measurement of surface electrocardiogram: the p-wave amplitude, P wave time duration and the p-wave duration dispersion (dP =Pmax- Pmin) of the same 12 lead electrocardiogram in the same cardiac cycle.Two cardiologists measured the value separately.The investigators record the mean value. 2). Atrial effective refractory period (AERP) measured from the high right atrium(HRA,the junction of superior vena cava and the right atrium , near the sinus node), low lateral right atrium(LLRA,the junction of inferior vena cava and the right atrium,on the right atrium free wall side), coronary sinus electrode (CS)7.8, and CS1.2 at 3 basic drive cycle lengths (CLs) of 600, 500, and 400 ms. Pacing was performed using a pulse width of 2 ms and a current output of twice the local diastolic threshold. If the latter was 2.0 milliampere (mA), the catheter was replaced and the threshold repeated. AERP was measured using an 8-beat drive train and a single extrastimulus incremented by 10 ms from a starting point of 170 ms. Every AERP was repeated 3 times, and the mean was taken. 3). At each CL, the dispersion of refractoriness was measured by subtracting the minimum from the maximum AERP across the 4 sites.
4. Rate adaption of AERP: With the gradual shortening of the pacing cycle lengths, the atrial effective refractory should be shortened accordingly. The rate adaption of AERP was observed in different pacing cycle lengths.
5. Atrial conduction time measured at the HRA after 30 seconds of constant pacing at a CL of 600, 500, and 400 ms. Conduction time is measured from the pacing artifact to the onset of the first initial sharp deflection recorded to the first A wave at CS1.10 and CS1.2. Total atrial conduction time=Pace HRA-Acs1.2; Right atrial conduction time=PaceHRA-Acs9.10; Left atrial conduction time=Acs9.10-Acs1.2.6). Atrial electromechanical conduction time: three sampling points are taken at lateral mitral valve(Sa1), septal mitral valve(Sa2), lateral tricuspid valve (Sa3), in the tissue doppler four-chamber view. Atrial electromechanical conduction time is measured from electrocardiogram P wave initiation to ultrasound A wave initiation. Total atrial electromechanical conduction time=T1-T3;Right atrial electromechanical conduction time=T2-T3; Light atrial electromechanical conduction time=T2-T1.

All patients fill the follow-up form before procedure. After catheter ablation therapy, all patients invited to come back to the outpatient clinic every week in the first month, and then at 2, 3, 6, 9, and 12 month to follow up. Patients received electrocardiogram and Holter monitor examination if with symptoms of palpitations. Those patients with no symptoms received electrocardiogram every month and Holter monitor examination every 6 months. Recurrence of atrial fibrillation was defined as atrial fibrillation/flutter or atrial tachycardia lasting ≥ 30 seconds 3 months after radiofrequency catheter ablation therapy. Patients who have AF recurrence within three months after therapy will not be considered for repeated radiofrequency ablation.Blood samples (routine blood, high sensitivity c-reactive protein,B-type natriuretic peptide (BNP), cystatin C,homocysteine,β2-microglobulin) and transthoracic echocardiography indexes (left atrial anterior to posterior diameter, left atrial length-diameter,left atrial transverse-diameter,left atrial volume index, mitral e', E peak, A peak, E/A,velocity time integral (VTI), left atrial ejection fraction, left atrial strain, strain rate and atrial electrical - mechanical conduction time) are recorded in all patients at each follow-up. Patients with AF recurrence must have an electrocardiogram or a 24 hour holter monitor evidence.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal AF episode occurs in the patient at least twice within half a year (electrocardiogram data or Holter), AF cannot be prevented in patients who orally take class I and III antiarrhythmic drugs, and patient age is ≤80 years.

Exclusion Criteria:

* patients with previous history of AF ablation, atrial thrombosis, or valvular heart disease (moderate and severe valvular stenosis, severe valvular regurgitation), left atrium (LA) >50 mm, patients who underwent prosthetic heart valve replacement, pregnant women, patients with existing liver and kidney disease, malignant tumors or hematological system diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change of P wave | 1-12 month
  Electrocardiogram
Atrial effective refractory period | During the operation
  Electrophysiological examination

SECONDARY OUTCOMES:
Plasma biomarkers of inflammation assessed | 1-12 month
  Blood samples are extracted in all patients for the detection of routine blood, high sensitivity c-reactive protein in mg/L,cystatin C in mg/L.
B type natriuretic peptide assessed | 1-12 month
  Blood samples are extracted in all patients to detected
Left atrial function | 1-12month
  Transthoracic echocardiography
Coagulation index assessed | 1-6 month
  Blood samples are extracted in all patients to detected
homocysteine assessed | 1-12 month
  Blood samples are extracted in all patients to detected
β2-microglobulin assessed | 1-12 month
  Blood samples are extracted in all patients to detected

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China